CLINICAL TRIAL: NCT01268579
Title: A Pilot Study to Assess the Pharmacodynamic Effects of Ribavirin in Patients With Tonsil and/or Base of Tongue Squamous Cell Carcinoma
Brief Title: Pharmacodynamic Effects of Ribavirin in Patients With Tonsil and/or Base of Tongue Squamous Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-218
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Results first posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-04

CONDITIONS: HEAD & NECK Cancer
Keywords: ribavirin; VIRAZOLE; tonsil; base of tongue; squamous cell carcinoma; 10-218
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Ribavirin

ARMS (1):
- ribavirin (Experimental): This will be a single institution non-randomized study for patients with tonsil and/or base of tongue squamous cell cancer. This is a pilot study to obtain pharmacodynamic data regarding the effects of ribavirin on tonsil squamous cell cancer.
  Interventions: Drug: ribavirin

INTERVENTIONS:
Drug: ribavirin — The clinical intervention in this study is ribavirin therapy for approximately 14 days. Ribavirin 800 mg/day is administered in divided doses, 400 mg PO qAM and 400 mg PO qPM.

SUMMARY:
Human papillomavirus (HPV-16) is an important factor in the development of many tonsil and/or base of tongue squamous cell cancers. Although HPV-16 is not thought to cause cancer by itself, it appears to contribute to the development of tonsil and/or base of tongue cancer in many patients. It is likely that treatment for many patients with tonsil and/or base of tongue cancer could be improved if effective therapy to control HPV-16 is developed. The investigators in this study want to learn if ribavirin shows evidence of activity against HPV-16.

Ribavirin is a pill therapy that is approved by the Food and Drug Administration (FDA) as part of the standard treatment for Hepatitis C. Laboratory experiments suggest that ribavirin might also be useful in the treatment of head and neck cancers. However, ribavirin has not yet been tested against head and neck cancer in patients. The purpose of this study is to find out the effects of ribavirin on tonsil and base tongue squamous cell cancer in patients.

The main purpose of this study is to see if ribavirin changes the expression of certain proteins related to HPV infection in the tumor. The study will also find out if ribavirin changes how the tumor appears in a PET/CT scan (positron emission tomography/computed tomography scan).

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnostic surgical or core needle biopsy, with confirmation of tonsil and/or base of tongue squamous cell carcinoma that is positive for expression of p16 and phosphorylated eIF4E, as determined by the Department of Pathology at MSKCC. The biopsy may be either of the tonsil base of tongue and/or an involved neck node. 2 unstained slides and/or tissue block must be available from the initial diagnostic biopsy
* Positive expression p16 and phosphorylated eIF4E is defined as >=30% of tumor cells with cytological and/or nuclear staining
* Age ≥ 18 and ≤ 65 years of age
* Karnofsky Performance Status ≥ 80
* Adequate organ function, as follows:

Adequate bone marrow reserve: absolute neutrophil count (ANC) ≥ 1.5 X 109/L, platelets ≥ 160 X 109/L, hemoglobin ≥ 12 g/dL Hepatic: total bilirubin within 1.5 X upper limit of normal (ULN) ; alkaline phosphatase (AP), aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 X ULN (Patients with Gilbert's syndrome as the cause of hyperbilirubinemia may be eligible if total bilirubin ≤ 2.5 X UNL) Renal: Serum creatinine ≤ 1.3 mg/dL. Patients with serum creatinine > 1.3 mg/dL may be eligible if creatinine clearance (CrCl) ≥ 55 mL/min based on the standard Cockroft and Gault formula.

* Patients of childbearing potential must have a negative serum pregnancy test within 14 days of treatment. Patients must agree to use a reliable method of birth control during and for 6 months following the last dose of study drug.
* Ability to swallow oral medication.
* Non-surgical patients: If primary radiation +/- chemotherapy (concurrent or sequential) is planned, patients must agree to undergo research biopsy after completion of ribavirin treatment.

Exclusion Criteria:

* Prior chemotherapy or radiation for tonsillar or base of tongue squamous cell cancer
* More than 10 pack-years of tobacco use
* History of hemolytic anemia or thalassemia
* Active infection or serious underlying medical condition that would impair the patient's ability to receive protocol treatment.
* Current therapeutic anticoagulation with Coumadin (warfarin)
* Current or prior treatment with ribavirin
* Known active Hepatitis B or C
* Any prior documented history of transient ischemic attack (TIA) or cerebrovascular accident (CVA)
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* Clinically significant peripheral vascular disease
* History of unstable angina or myocardial infarction (MI) within the last 3 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-12-28 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Pfisher, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Burman B, Drutman SB, Fury MG, Wong RJ, Katabi N, Ho AL, Pfister DG. Pharmacodynamic and therapeutic pilot studies of single-agent ribavirin in patients with human papillomavirus-related malignancies. Oral Oncol. 2022 May;128:105806. doi: 10.1016/j.oraloncology.2022.105806. Epub 2022 Mar 23. PMID 35339025
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ribavirin
Started | 9
Completed | 6
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ribavirin
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 59 [47 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: To Explore if Ribavirin Therapy for 2 Weeks Decreases Tumor Expression
Description: of phosphorylated eIF4E among patients with tonsillar squamous cell carcinoma.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ribavirin
Number analyzed (Participants) | 9
Participants
  Decreased p-eIF4E after 14 days of ribavirin | 4
  No decreased p-eIF4E after 14 days of ribavirin | 2
  Not evaluable | 3

2. Secondary Outcome: to Explore the Pharmacodynamic Effects of Ribavirin
Description: on molecules that may be regulated directly or indirectly by eIF4E (eg, p16, p21, EGFR, p53).). Immunohistochemistry will be performed on Pathology samples (e.g. diagnostic biopsy), as well as on the post-treatment surgical pathology samples (e.g. definitive surgery),to describe the effects of ribavirin treatment on the expression of phosphorylated eIF4E.
Time Frame: pre-treatment and post treatment
Population: N/A - data were not collected
Arm/Group | Ribavirin
Number analyzed (Participants) | 0

3. Secondary Outcome: To Explore if Ribavirin Reduces the Expression of HPV-16 Oncoproteins E6 and E7
Description: Pathology samples (e.g. diagnostic biopsy), as well as on the post-treatment surgical pathology samples (e.g. definitive surgery)
Time Frame: In pre- and post-treatment tumor samples
Population: N/A - data were not collected
Arm/Group | Ribavirin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Ribavirin
All-Cause Mortality (participants affected / at risk) | 8/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ribavirin (N=9)
Anemia (Blood and lymphatic system disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Blood bilirubin increase (Investigations) | 3
Fatigue (General disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Aspartate aminotransferase increase (Investigations) | 2
Fever (General disorders) | 2
Gastroesophageal Reflux (Gastrointestinal disorders) | 2
Weight loss (Investigations) | 2
Alanine aminotransferase increase (Investigations) | 1
Alkaline phosphatase increase (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT01268579/Prot_SAP_000.pdf